CLINICAL TRIAL: NCT05640375
Title: Comparison of Follow-up and Steroid Treatment Results in Intussusception in Children
Brief Title: Follow-up and Steroid Treatment Results in Intussusception
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Tuğba Acer Demir, Clinical Associate Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUTF-TAcerDemir-001
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Intussusception
Keywords: Intussusception; steroid; methylprednisolone
MeSH Terms: conditions — Intussusception | interventions — Methylprednisolone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow-up (No Intervention): Intussuception diagnosed, Informed consent was obtained by explaining treatment options to their families, no tenderness on abdominal examination, the duration of complaints is less than 24 hours, no findings of complication, Just IV hydration and ultrasonography is repeated 4 hours later (clinical and physical examination findings are monitored)
- Single dose Steroid treatment (Experimental): Intussuception diagnosed, Informed consent was obtained by explaining treatment options to their families, no tenderness on abdominal examination, the duration of complaints is less than 24 hours, no findings of complication, Methylprednisolone 1 mg/ kg single dose was given and ultrasonography is repeated 4 hours later (clinical and physical examination findings are monitored)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Single dose, 1 mg/kg
  Other Names: Steroid
  Arms: Single dose Steroid treatment

SUMMARY:
Treatment interventions in the treatment of intussusception are hydrostatic or pneumatic reduction and manual reduction with laparotomy. In addition, it is known that in some of the ileoileal intussusception cases, intussusception disappears in short-term observation and it is an accepted treatment to follow-up for a while in ileoileal cases without making a decision for laparotomy. In a study the investigators conducted, they reported that 17 of 81 patients had spontaneous opening with follow-up and no further treatment was required. The hydrostatic or pneumatic reduction has a 0.8% risk of bowel perforation, fever due to bacterial translocation is common, septicemia has also been reported and anal fissures due to catheterization is seen. Baby or child's stress, psychology, abdominal pain are other negative aspects that cannot be measured. In a study that was reported a patient with HSP was diagnosed with intussusception while under steroid treatment, and when the patient was taken to laparoscopy, it was observed that the patient's intussusception was opened. In the same study, the authors mentioned that they followed up 4 patients diagnosed with HSP by administering only steroid treatment and observed that intussusception was opened in 3 of these patients without the need for any other intervention.

The steroid is used as a single dose (1 mg/kg) in cases such as acute allergic reactions, bronchiolitis, asthma, laryngitis, edema treatment, bronchoscopy, intubation, extubation medication. When the literature is reviewed, it has been shown that single-dose, low-amount (1 mg/kg) steroid therapy does not have side effects. The investigators predict that the steroid will reduce the thickening of Peyer's plaques with its anti-inflammatory effect, and relieve edema as in other areas of use, by relieving the congested intussusceptum. Thus, in infants and children, there will be no need for hydrostatic or pneumatic reduction, which has the risk of perforation and infection (septicemia) and exposure to radiation, and our patients will regain their health without the need to apply this interventional treatment.

DETAILED DESCRIPTION:
Treatment interventions in the treatment of intussusception are hydrostatic or pneumatic reduction and manual reduction with laparotomy. In addition, it is known that in some of the ileoileal intussusception cases that cannot be reached with hydrostatic or pneumatic reduction, intussusception disappears in short-term observation and control ultrasound (USG), and it is an accepted treatment to follow-up for a while in ileoileal cases without making a decision for laparotomy. In a study the investigators conducted, they reported that 17 of 81 patients had spontaneous opening with follow-up and no further treatment was required.

In hydrostatic or pneumatic reduction, a catheter is inserted into the rectum from the anus of the infant or child patient, and the catheter balloon is inflated in a way that does not allow liquid or gas escape. Afterwards, barium, saline (SF) or air is given through this probe with limited pressure (limited pressure is given due to the risk of bowel perforation), the patient is tried to be kept still and an image is taken under fluoroscopy, or if there is an experienced radiologist, SF is given, followed by USG. This procedure has a 0.8% risk of bowel perforation. At the same time, fever due to bacterial translocation is common, septicemia has also been reported. Anal fissures due to catheterization are tried to be treated with warm water pad application after the procedure. Since the follow-up of the procedure is carried out under the scope, the patients are also exposed to radiation. Baby or child's stress, psychology, abdominal pain are other negative aspects that cannot be measured.

As another treatment, surgery includes negative effects such as leaving a scar on the skin, exposing the patient to the risk of adhesion and intestinal obstruction due to adhesion, risk of anesthesia as a surgical procedure, and risk of bleeding and infection.

In a study that was reported a patient with HSP was diagnosed with intussusception while under steroid treatment, and when the patient was taken to laparoscopy, it was observed that the patient's intussusception was opened. In the same study, the authors mentioned that they followed up 4 patients diagnosed with HSP by administering only steroid treatment and observed that intussusception was opened in 3 of these patients without the need for any other intervention. In another study a case of intussusception that recurred 9 times was reported and after investigating the underlying cause, the authors found that the only cause was lymphoid hyperplasia, and they reported that intussusception did not recur after steroid treatment was applied to this patient. . In another study, the authors did not detect any cause other than lymphoid hyperplasia in two cases with recurrent intussusception and that success was achieved with steroid treatment. Although it has been reported that the use of steroid therapy together with hydrostatic or pneumatic reduction causes recurrence at a lower rate than the patients who received only hydrostatic or pneumatic reduction therapy, a study found no difference in this direction.

95% of intussusceptions are idiopathic. In these patients, intussusception is thought to be caused by Peyer's plaques (lymphoid tissue in the intestinal wall) thickened in response to an infection. The increase in the frequency of intussusception after rotavirus vaccine supports this idea.

The steroid is used as a single dose (1 mg/kg) in cases such as acute allergic reactions, bronchiolitis, asthma, laryngitis, edema treatment, bronchoscopy, intubation, extubation medication. When the literature is reviewed, it has been shown that although chronic and high-dose steroid therapy has side effects, single-dose, low-amount (1 mg/kg) steroid therapy does not have side effects. It is seen that this treatment, which is used when necessary in patients presenting to the emergency department, is used alone in HSP patients in patients with intussusception, and in combination with hydrostatic or pneumatic reduction after treatment in recurrent intussusception cases, to prevent recurrence and to reduce the risk of recurrence.

Recently, with the frequent use of USG, the diagnosis of intussusception is made early and in large numbers, and the prognosis of intussusceptions that are caught early is better. When the investigators examined their cases in the last 10 years, the investigators found that 80% of their cases were diagnosed with a complaint period of less than 24 hours.

The investigators predict that the steroid will reduce the thickening of Peyer's plaques with its anti-inflammatory effect, and relieve edema as in other areas of use, by relieving the congested intussusceptum. Thus, in infants and children, there will be no need for hydrostatic or pneumatic reduction, which has the risk of perforation and infection (septicemia) and exposure to radiation, and our patients will regain their health without the need to apply this interventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* who applied to Başkent University Ankara Hospital Pediatric Emergency Polyclinic,
* Diagnosed with intussusception by USG,
* Consulted with Pediatric Surgery
* Informed consent was obtained by explaining treatment options to their families.

Exclusion Criteria:

* Diffuse tenderness and defense on abdominal examination,
* The duration of the complaints exceeds 24 hours,
* When the intestinal blood supply is decreased in the ultrasound findings,
* Patients with free air on the standing abdominal X-ray,
* Patients with pathology requiring urgent surgical intervention

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Treatment of intussusception | 4 hours later
  Ratio of Participants with No intussusception on ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Ender Fakıoğlu, Principal Investigator — Baskent Univesity
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD can be shared if a colleague needs and wants after the article is published

REFERENCES:
- [Derived] Acer-Demir T, Gultekingil A, Fakioglu E, Guney LH, Sezer R. Successful Treatment of Early Presenting Intussusception With a Single Dose of Corticosteroid: A Prospective Randomized Controlled Trial. J Pediatr Surg. 2025 Apr;60(4):162198. doi: 10.1016/j.jpedsurg.2025.162198. Epub 2025 Jan 25. PMID 39914152